CLINICAL TRIAL: NCT07381933
Title: The Effect of Consumed Berries on Extracellular Vesicle Signalling in the Body
Acronym: NutriEV RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Collaborators: European Innovation Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2025-16589; 101161353 (Other Grant/Funding Number: European Innovation Council (EIC))
Record Dates: First submitted 2025-09-30; First posted 2026-02-02 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Healthy; Extracellular Vesicles
Keywords: extracellular vesicles

STUDY DESIGN:
Intervention Model Description: Participants are randomized (using block randomization) into two groups. Each group receives a different intervention (cloudberries or lingonberries). Both groups are treated simultaneously (in parallel) The design compares outcomes between these two parallel arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cloudberry Group (Experimental): 30 participants will be allocated to Cloudberry Group.
  Interventions: Dietary Supplement: Cloudberries
- Lingonberry Group (Experimental): 30 participants will be allocated to Lingonberry Group.
  Interventions: Dietary Supplement: Lingonberries

INTERVENTIONS:
Dietary Supplement: Cloudberries — Participants consume 270 grams (equivalent of 3 dl) of cloudberries orally twice daily for 7 days.
  Arms: Cloudberry Group
Dietary Supplement: Lingonberries — Participants consume 200 grams (equivalent of 3 dl) of lingonberries orally twice daily for 7 days
  Arms: Lingonberry Group

SUMMARY:
This study examines how berry consumption influences the signaling and distribution of extracellular vesicles (EVs) in the human body. EVs are small bilipid-layered nanoparticles released by cells. EVs carry proteins, lipids, and genetic material, and play a key role in cell-to-cell communication. The composition of EVs reflects the state of their cells of origin, and EVs can affect other cells by delivering their biological contents. EVs offer significant potential for both diagnostics and new therapies.

Recent research has shown that EVs can be found in blood, urine, sweat, and can even cross biological barriers such as the blood-brain barrier and placenta. Many living organisms, including mammalian cells, bacteria, and plants, release EVs. Berries such as cloudberries and lingonberries have demonstrated positive effects on gut microbiota and metabolism, supporting digestive and metabolic health.

In this study, a nutritional intervention will be conducted to investigate the effects of berry consumption on extracellular vesicle signaling of human cells and the gut microbiota, as well as the biodistribution of berry-derived vesicles in the human body.

DETAILED DESCRIPTION:
This randomized clinical pilot study will enroll 60 healthy adults. Participants will consume either 270 grams of cloudberries or 200 grams of lingonberries (equivalent of 3 dl) daily, for 7 days.

Urine, sweat and faecal samples will be collected from participants both before and after the nutritional intervention. Researchers will isolate EVs from samples and analyze the isolated EVs using transmission electron microscopy (TEM), 16S RNA sequencing, proteomics, and metabolomics. The results obtained from vesicle analyses before and after the nutritional intervention will be compared. Additionally, blood samples will be collected to monitor the immunological status of participants and also information on participants' dietary habits will be collected through a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50
* Individuals of all heights and weights and both female and male sexes are accepted
* Written informed consent is required from all study participants
* Use of probiotics is allowed, but the usage will be reported

Exclusion Criteria:

* Known or suspected allergy to cloudberries or lingonberries
* Current dermatological or gastrointestinal conditions requiring treatment or interfering the sampling
* Renal failure
* Type 1 or type 2 diabetes
* Pregnancy
* Immunodeficiency or any condition affecting the immune system, e.g. chronic viral infection
* Ongoing antibiotic treatment or antibiotic treatment within the past 3 months
* Immunosuppressive medication or other medication that can be influenced by the intervention

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-23 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Impact of Dietary Berries on Extracellular Vesicle Communication and Host Immunity | From baseline (pre-intervention) to Day 7 (post-intervention)
  The investigators will assess the effects of berry consumption on the human body, including alterations in gut microbiota composition and immune cell profiles, with a particular focus on changes in extracellular vesicle (EV) signaling.

SECONDARY OUTCOMES:
Changes in Plasma Cytokine Profiles Following Dietary Intervention | Baseline (pre-intervention) to Day 7 (post-intervention)
  The investigators will quantify plasma cytokine levels (e.g. IL-6, TNF-α, IL-10) from the participants' blood samples to assess systemic immunological response to the dietary intervention.
Host Response in Blood Following Dietary Intervention | Baseline (pre-intervention) to Day 7 (post-intervention)
  The investigators will analyse host immunological response to the dietary intervention via blood sample analysis. Peripheral white blood cell subsets (e.g. T cells, B cells and monocytes) will be determined using flow cytometry to evaluate cellular immune response.
Detection and quantification of Berry-Derived Extracellular Vesicles in Human Faeces | From baseline to Day 7 (post-intervention)
  The investigators will detect the presence of the berry-derived EVs in faeces after a dietary intervention.
Detection and Quantification of Berry-Derived Extracellular Vesicles in Human Urine | From baseline to Day 7 (post-intervention)
  The investigators will detect the presence of the berry-derived EVs outside the intestinal tract in urine after a dietary intervention.
Detection and Quantification of Berry-Derived Extracellular Vesicles in Human Sweat | From baseline to Day 7 (post-intervention)
  The investigators will detect the presence of the berry-derived EVs outside the intestinal tract in sweat after a dietary intervention.
Changes in Extracellular Vesicle Size, Concentration, and Cargo after Nutritional Intervention | From baseline (pre-intervention) to Day 7 (post-intervention)
  The investigators will detect changes in EV properties such as size, concentration, and cargo profile following the dietary intervention, when analysing urine, faecal and sweat samples before and after the dietary intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Oulu University Hospital, Oulu, Finland

IPD SHARING:
Plan to Share IPD: No
IPD will be shared after reasonable request

REFERENCES:
- See also: NutriEV project website — https://nutrievproject.eu/